# **Study Documents**

# **Cover Page**

**Official Title of the study:** An Exploratory Study on the Impact of Prolonged Postoperative Endotracheal Extubation Time on Postoperative Complications in Gastric Cancer Patients with Severe Obstructive Sleep Apnea

**NCT number:** NCT ID not yet assigned

Date of the document: 2026.1.15

**Official Title of the study:** An Exploratory Study on the Impact of Prolonged Postoperative Endotracheal Extubation Time on Postoperative Complications in Gastric Cancer Patients with Severe Obstructive Sleep Apnea

NCT number: NCT ID not yet assigned Unique Protocol Id: KYLL-202110-034-2

Date of the document: 2026.1.15

# **Clinical Study Protocol**

**Project Title:** An Exploratory Study on the Impact of Prolonged Postoperative Endotracheal Extubation Time on Postoperative Complications in Gastric Cancer Patients with Severe Obstructive Sleep Apnea

**Research Unit:** <u>Department of General Surgery, Qilu Hospital of Shandong University</u>

**Principal Investigator:** <u>Yu Wenbin</u>

**Sponsor:** <u>Qilu Hospital of Shandong University</u>

# **Study Abstract**

| Item | Content |
|---|---|
| Project Title | An Exploratory Study on the Impact of Prolonged<br>Postoperative Endotracheal Extubation Time on<br>Postoperative Complications in Gastric Cancer<br>Patients with Severe Obstructive Sleep Apnea |
| Study Objective | To investigate the impact of prolonging the time to postoperative endotracheal extubation on the incidence of postoperative complications in gastric cancer patients with severe obstructive sleep apnea. |
| Research<br>Hypothesis | Prolonging the time to endotracheal extubation in gastric cancer patients with severe obstructive sleep apnea can reduce the incidence of postoperative complications. |
| Study Design | □ Case-Control Study 🗷 Cohort Study □ |

Item Content

Cross-Sectional Study

☐ Case Report / Case Series

#### Inclusion Criteria:

- 1. Patients preoperatively diagnosed with resectable gastric cancer.
- 2. Patients without distant organ metastasis.
- 3. Patients with preoperative OCST or PSG results showing AHI >30 events/hour and  $SaO_2 < 80\%$ .
- 4. Patients with cardiopulmonary function deemed suitable for surgery.
- 5. Patients aged 18-85 years.
- 6. Patients who voluntarily joined this study and provided written informed consent.

## Exclusion Criteria:

# Study Subjects

- 1. Patients with a history of or concurrent other malignant tumors.
- 2. Patients who underwent palliative resection.
- 3. Subjects who experienced acute cardiovascular or cerebrovascular events (e.g., acute cerebral infarction, acute coronary syndrome) within the past 3 months, or whose cardiovascular clinical symptoms/diseases are not well-controlled.
- 4. Patients with a history of psychotropic drug abuse that cannot be abstained, or those with psychiatric disorders.
- 5. Patients with concomitant diseases that, in the investigator's judgment, seriously endanger the patient's safety or affect the completion of the study.

Meet either (A + B) or C below.

A: Presence of at least 1 of the following: (1) Patient complaints of sleepiness, non-restorative sleep, fatigue, or insomnia; (2) Waking from sleep due to choking or gasping; (3) Bed partner or other observer reports of habitual snoring, breathing interruptions, or both during sleep; (4) Diagnosed hypertension, mood disorder, cognitive dysfunction, coronary artery disease, cerebrovascular disease, congestive heart failure, atrial fibrillation, or type 2 diabetes.

B: PSG or OCST confirms ≥5 respiratory events/hour during monitoring, including obstructive apneas,

# Diagnostic Criteria

Item Content

mixed apneas, hypopneas, and respiratory effort-related arousals (RERAs).

C: PSG or OCST confirms ≥15 respiratory events/hour during monitoring, including obstructive apneas, mixed apneas, hypopneas, and RERAs.

The incidence of postoperative complications in gastric cancer patients with severe sleep apnea is the primary endpoint of this study. Based on previous large-scale literature reports, the incidence of perioperative cardiovascular complications in patients with severe sleep apnea undergoing non-cardiac surgery is 15% higher than in the normal population [8]. Using a power of 90% and a significance level of 5%, sample size estimation was performed using PASS, version 11 (NCSS, LLC). We need to recruit 93 patients per group. Accounting for loss to follow-up, dropouts, and other factors, we plan to include at least 120 patients per group.

Sample Size & Justification

Primary Exposure Factor

Time to endotracheal extubation

Outcome Variables

Incidence of short-term postoperative complications, graded using the Clavien-Dindo classification.

Follow-up Plan (For Cohort Studies) Routine follow-up examinations at 1, 3, 6, 9, and 12 months postoperatively. Collect routine follow-up indicators and assess the occurrence of postoperative complications.

Sample Collection

☑ No ☐ Yes

Brief description of tissue type and quantity: N/A

Non-Medical Purpose

Examinations

☑ No □ Yes

e.g., unnecessary CT scans, contrast studies, lab tests, etc.: N/A

Statistical Methods Chi-square test or Fisher's exact test will be used to compare categorical variables. Continuous variables will be expressed as median and IQR if non-normally distributed and analyzed using the Mann-Whitney U test, or as mean (SD) if normally distributed and analyzed using the t-test.

Study Risk
Self-Assessment

□ High-Risk Study □ Medium-Risk Study ☑ Low-Risk Study

Brief explanation: This is an observational study.

# Confidentiality Statement:

The information contained in this study protocol is provided solely to the investigators of this project, the clinical research management committee, and relevant regulatory bodies for review. Disclosing any information to third parties unrelated to this study is strictly prohibited without the approval of the Principal Investigator.

# 1. Research Background (State the rationale and significance of this study based on current domestic and international research)

As one of the most common malignant tumors worldwide, gastric cancer ranks fifth in global cancer incidence and fourth in cancer mortality [1]. Current treatment for gastric cancer is comprehensive, primarily based on surgical treatment, with standard radical gastrectomy being the main procedure [2]. This process is complex, technically demanding, and carries relatively high surgical risks. Obstructive Sleep Apnea (OSA) is a sleep-related breathing disorder characterized by periodic partial or complete upper airway obstruction during sleep, manifesting as apneas and hypopneas [3]. Preliminary statistics indicate the overall prevalence of OSA among adults in China is 3.93% [4], yet the clinical diagnosis rate remains low. OSA is widely recognized as an independent risk factor for hypertension and metabolic syndrome [5, 6]. Reported prevalence of OSA among surgical patients is approximately 7%-10%, but can reach 68%-70% in high-risk populations (bariatric surgery or other major non-cardiac surgery). These patients have significantly increased perioperative complications and mortality [7, 8], especially severe sleep apnea. One cohort study reported the incidence of cardiovascular complications within 30 days after surgery in patients with severe sleep apnea was as high as 30.1% [8]. General anesthesia, sedatives, and postoperative analgesics are potent respiratory depressants; they can relax the upper airway dilator muscles and impair the ventilatory response to hypoxemia and hypercapnia. These effects exacerbate OSA. Concurrently, the hypoxemia caused by OSA can increase the incidence of postoperative complications in gastric cancer patients and may predispose them to postoperative cardiovascular complications [9]. Therefore, for gastric cancer patients with severe sleep apnea, strategies to reduce postoperative complications and adverse events are particularly important.

# 2. Research Question & Objectives (Elucidate the scientific question and research objectives)

To investigate the impact of prolonging the time to postoperative endotracheal extubation on the incidence of postoperative complications in gastric cancer patients with severe obstructive sleep apnea.

#### 3. Research Methods (This section should be elaborated in detail)

## **Study Design**

This is a single-center, prospective cohort study. Starting June 2025, the study plans to enroll patients undergoing radical gastrectomy for gastric cancer in the Department of General Surgery of our hospital who also have severe obstructive sleep apnea. Based on the anesthesiologist's assessment during the perioperative period regarding sufficient metabolism of anesthetic agents and full patient awakening, patients will be divided into two groups regarding whether extubation time is prolonged (by 1-2 days): Exposure Group: Prolonged extubation time group; Non-Exposure Group: Non-prolonged extubation time group (extubation on the day of surgery group). Clinical data, intraoperative details, postoperative pathology, lymph node status, and postoperative complications will be recorded for all patients.

# Study Site and Subjects (Source, Inclusion, and Exclusion Criteria)

All patients in this study will be inpatients from the Department of Gastrointestinal Surgery, Qilu Hospital.

#### **Inclusion Criteria:**

Patients preoperatively diagnosed with resectable gastric cancer.

Patients without distant organ metastasis.

Patients with preoperative OCST or PSG results showing AHI >30 events/hour and  $SaO_2 < 80\%$ .

Patients with cardiopulmonary function deemed suitable for surgery.

Patients aged 18-85 years.

Patients who voluntarily joined this study and provided written informed consent.

#### **Exclusion Criteria:**

Patients with a history of or concurrent other malignant tumors.

Patients who underwent palliative resection.

Subjects who experienced acute cardiovascular or cerebrovascular events (e.g., acute cerebral infarction, acute coronary syndrome) within the past 3 months, or whose cardiovascular clinical symptoms/diseases are not well-controlled.

Patients with a history of psychotropic drug abuse that cannot be abstained, or those with psychiatric disorders.

Patients with concomitant diseases that, in the investigator's judgment, seriously endanger the patient's safety or affect the completion of the study.

# **Study Variables (Factors) and Measurement**

Study Variable: Whether endotracheal extubation time is prolonged.

# **Study Outcomes**

Incidence of short-term postoperative complications, graded using the Clavien-Dindo classification.

# Follow-up (For Cohort Studies)

Routine follow-up examinations at 1, 3, 6, 9, and 12 months postoperatively. Collect routine follow-up indicators and assess the occurrence of postoperative complications.

# Sample Size

The incidence of postoperative complications in gastric cancer patients with severe sleep apnea is the primary endpoint of this study. Based on previous large-scale literature reports, the incidence of perioperative cardiovascular complications in patients with severe sleep apnea undergoing non-cardiac surgery is 15% higher than in the normal population [8]. Using a power of 90% and a significance level of 5%, sample size estimation was performed using PASS, version 11 (NCSS, LLC). We need to recruit 93 patients per group. Accounting for loss to follow-up, dropouts, and other factors, we plan to include 120 patients per group, totaling an estimated 240 patients for both groups.

# **Study Flowchart**

Gastric cancer patients with severe sleep apnea

- -> Apply Inclusion/Exclusion Criteria
- -> Undergo surgical treatment
- -> Decision on prolonging extubation time?

```
text
```

```
Yes -> Exposure Group: Prolonged extubation time text
```

No -> Non-Exposure Group: Non-prolonged extubation time

Compare complication rates between the two groups

- -> Follow-up for 1 year
- -> Compare complication rates between the two groups

## **Data Collection and Management**

Preoperative patient status: General information (name, gender, age, BMI),

preoperative nutritional status, preoperative tumor marker levels, preoperative comorbidities, etc.

Postoperative recovery: Time to recovery of bowel function (first flatus, first oral water/fluid intake), postoperative complications (pulmonary infection, postoperative gastroparesis, postoperative reflux, inflammatory bowel obstruction, bleeding, perforation, anastomosis-related complications such as anastomotic leak, anastomotic stenosis, anastomotic bleeding, etc.), cardiovascular and cerebrovascular complications, etc.

Postoperative follow-up information: Patient review at 1, 3, 6, 9, and 12 months postoperatively, CT and gastroscopy results.

## **Statistical Analysis Methods**

Chi-square test or Fisher's exact test will be used to compare categorical variables. Continuous variables will be expressed as median and IQR if non-normally distributed and analyzed using the Mann-Whitney U test, or as mean (SD) if normally distributed and analyzed using the t-test. Survival data will be analyzed using Kaplan-Meier curves. Enrollment is expected to be completed between June 2025 and June 2026. Follow-up is expected to be completed between June 2026 and June 2027.

# **Quality Control**

During the clinical research process, strictly adhere to the procedures specified in the clinical study protocol. Collect and enter data completely and accurately. Manage data using a standardized database.

# 4. Feasibility Analysis

This is an observational study requiring no additional medical procedures or expenses, making it technically and economically feasible.

## 5. Timeline

Enrollment is expected from June 2025 to June 2026.

Follow-up is expected from June 2026 to June 2027.

Data analysis and manuscript writing are expected to be completed by December 2027.

# 6. References

- Sung HA-O, Ferlay J, Siegel RA-O, Laversanne M, Soerjomataram I, Jemal A, Bray F: Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. (1542-4863 (Electronic)).
- 2. Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition). (1436-3305 (Electronic)).
- 3. 陈裕桦, 高媛, 王连城, 郭子煜, 付善民: **成人阻塞性睡眠呼吸暂停治疗研究进展**. *临床口腔医学杂志* 2023, **39**(03):186-189.
- 4. 潘悦达, 王东博, 韩德民: 我国成人阻塞性睡眠呼吸暂停低通气综合征患病率的

- Meta 分析. 医学信息 2019, **32**(07):73-77+81.
- 5. Cadby G, McArdle N, Briffa T, Hillman DR, Simpson L, Knuiman M, Hung J: **Severity of OSA** is an independent predictor of incident atrial fibrillation hospitalization in a large sleep-clinic cohort. (1931-3543 (Electronic)).
- 6. Hirotsu C, Haba-Rubio J, Togeiro SM, Marques-Vidal P, Drager LF, Vollenweider P, Waeber G, Bittencourt L, Tufik S, Heinzer R: Obstructive sleep apnoea as a risk factor for incident metabolic syndrome: a joined Episono and HypnoLaus prospective cohorts study. LID 1801150 [pii] LID 10.1183/13993003.01150-2018 [doi]. (1399-3003 (Electronic)).
- 7. Hallowell PT, Stellato Ta Fau Schuster M, Schuster M Fau Graf K, Graf K Fau Robinson A, Robinson A Fau Crouse C, Crouse C Fau Jasper JJ, Jasper JJ: **Potentially life-threatening sleep apnea is unrecognized without aggressive evaluation**. (1879-1883 (Electronic)).
- 8. Chan MTV, Wang CY, Seet E, Tam S, Lai HY, Chew EFF, Wu WKK, Cheng BCP, Lam CKM, Short TG et al: Association of Unrecognized Obstructive Sleep Apnea With Postoperative Cardiovascular Events in Patients Undergoing Major Noncardiac Surgery. (1538-3598 (Electronic)).
- 9. Subramani Y, Singh M Fau Wong J, Wong J Fau Kushida CA, Kushida Ca Fau Malhotra A, Malhotra A Fau Chung F, Chung F: **Understanding Phenotypes of Obstructive Sleep Apnea: Applications in Anesthesia, Surgery, and Perioperative Medicine**. (1526-7598 (Electronic)).

Filename: 9. Study Protocol v1.5 2025.6.16.docx